CLINICAL TRIAL: NCT05586854
Title: Multicenter Study on Dialysis Modalities for End-stage Chronic Renal Failure Patients With Heparin-induced Thrombocytopenia
Acronym: MODIATIH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ramsay Générale de Santé (Other)
Collaborators: European Clinical Trial Experts Network (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-A00610-41
Record Dates: First submitted 2022-10-17; First posted 2022-10-19 (Actual); Last update posted 2022-10-19 (Actual); Status verified 2022-10

CONDITIONS: Dialysis; Complications; Heparin-induced Thrombocytopenia; Chronic Renal Failure
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Intervention Model Description: interventional, prospective, multicentre, longitudinal, non-comparative study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- end-stage renal disease patients with heparin-induced thrombocytopenia (Experimental): The research procedure consists of dialysing patients on a Hydrolink-NV® membrane with an anticoagulant dose decrease protocol. This protocol of decrease is done over a period of about 6 months divided into 4 periods.
  Interventions: Procedure: Hydrolink NV membrane

INTERVENTIONS:
Procedure: Hydrolink NV membrane — patient dialysis on a Hydrolink-NV® membrane with an anticoagulant dose decrease protocol.
  Period 1 : conventional membrane with his usual anticoagulant for 4 weeks. Period 2 : Hydrolink-NV® membrane with maintenance of the previous doses of Orgaran® Period 3 : Hydrolink-NV® membrane with a decrease in Orgaran® Period 4 : Hydrolink-NV® membrane with the minimum effective dose of Orgaran® or without Orgaran® for a period of 3 months (M4, M5, M6).

SUMMARY:
This research is based on the hypothesis that the Hydrolink®-NV dialysis membrane could allow the realization of quality dialysis with a significant reduction in the doses of Orgaran®, or even a total cessation of the anticoagulant, in patients with chronic renal failure. with heparin-induced thrombocytopenia.

Thus, this study aims to show that the use of this dialysis membrane without prior anticoagulation does not increase the risk of coagulation of the circuit and allows the realization of quality dialysis sessions.

ELIGIBILITY:
Inclusion Criteria:

* Patient, male or female, over 18 years of age.
* Patient on dialysis in a hemodialysis unit of the Ramsay Santé group.
* Patient with diagnosed heparin induced thrombocytopenia.
* Patient whose dialysis sessions benefit from extracorporeal circulation anticoagulation with Orgaran® or its equivalent (Arixtra® or Arganova®).
* Patient informed and having signed his written consent to participate in the study.
* Affiliated patient or beneficiary of a social security scheme.
* Woman of childbearing age with effective contraception, after verification of the absence of active pregnancy (negative pregnancy test)

Exclusion Criteria:

* Patient whose duration of dialysis is less than 1 month.
* Medically unstable or fragile patient.
* Patient participating in another clinical study.
* Protected patient: adult under guardianship, curatorship or other legal protection, deprived of freedom by judicial or administrative decision.
* Pregnant, breastfeeding or parturient women.
* Patient hospitalized without consent.
* Patient with severe hepatic failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-11-20 (Estimated); Primary Completion 2023-11-20 (Estimated); Study Completion 2024-06-20 (Estimated)

PRIMARY OUTCOMES:
The occurrence, or not, of a success of the dialytic technique. | 7 months
  The success of the dialytic technique is defined as the reduction, over the whole of period 4 of the study, of at least 50% of the dose of Orgaran® received by the patient at each dialysis session, compared to to that administered in period 2 of the study.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Privé Claude Galien, Quincy-sous-Sénart, France